CLINICAL TRIAL: NCT01399866
Title: Cognitive Remediation With D-cycloserine to Improve Smoking Cessation Outcomes
Brief Title: Cognitive Remediation With D-Cycloserine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, A. Eden Evins, Director Center for Addiction Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2011P000411
Record Dates: First submitted 2011-07-19; First posted 2011-07-22 (Estimated); Results first posted 2015-05-04 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-08

CONDITIONS: Smoking Cessation
Keywords: D-cycloserine; Smoking cues; Cognitive remediation; physiologic reactivity; craving
MeSH Terms: conditions — Smoking Cessation | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 50 mg capsule,single dose, twice, one week apart, by mouth
  Interventions: Drug: Placebo
- D-cycloserine (Active Comparator): 50 mg capsule,single dose, twice, one week apart, by mouth
  Interventions: Drug: D-cycloserine

INTERVENTIONS:
Drug: D-cycloserine — 2 single weekly doses, 50 mg capsule
  Arms: D-cycloserine
Drug: Placebo
  Arms: Placebo

SUMMARY:
One hundred seventy-five eligible participants will be enrolled with aim of randomizing 60 to a double-blind, placebo-controlled trial of D-cycloserine added to cue-exposure treatment to prevent relapse to smoking. Subjects who sign an informed consent, meet inclusion criteria, and demonstrate response to cue reactivity at the screening visit, will either be:

* started on approximately 3 weeks of either nicotine replacement therapy (NRT) at a dose of either 14 or 21 mg/day or varenicline titrated to 1.0 mg bid; decision of which method to use to quit smoking will be based on participant choice as well as taking into account any medical contraindications to either therapy.
* evaluated to confirm abstinence from smoking. Recently abstinent participants referred by a smoking cessation clinic, PCP or self referred must have an expired air CO < 10 ppm to confirm abstinence.

Subjects who are able to demonstrate 18-24 hours of abstinence prior to the first Cue Exposure Therapy Visit (CET I) will be eligible to be randomized to two visits of study medication and cue exposure treatment, spaced five to nine days apart. Subjects will complete 2 follow-up visits at 2-4 days and four weeks after the last CET visit. The entire study involves twelve visits and will last approximately ten weeks. For recently abstinent participants referred by a smoking cessation clinic, PCP or self referred, the study involves 7 visits (screening and baseline visit will be merged into one and there is no CBT component) and will last approximately 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have smoked an average of ≥ 10 cigarettes/day during the past 6 months
* have expired air CO ≥ 10 ppm or urine cotinine ≥ 100 ng/mL
* meet DSM-IV criteria for nicotine dependence
* aged 18 - 65
* Recently abstinent participants referred by a PCP, smoking cessation clinic or self referred must have an expired air CO < 10 ppm to confirm abstinence

Exclusion Criteria:

* Severe or uncontrolled medical or psychiatric illness
* History of multiple hospitalizations within the last six months for an ongoing medical condition
* Any significant, current and unstable cardiovascular disease, end stage renal failure, severe COPD requiring oxygen, any current unstable neurological disease, a history of seizures or epilepsy, or a history of head trauma with lasting neurological sequelae, will be excluded for their safety.
* Major depressive episode, mania or mixed episode in the prior 6 months
* Lifetime history of psychosis, delusional disorder, organic mental disorder by DSM-IV criteria, or ongoing cognitive impairment will also be excluded for their safety,
* Current excessive use of alcohol (>21 drinks/week in female subjects; >28 drinks/week in male subjects)
* Current use of illicit drugs.
* Current steroid use, current, daily use of benzodiazepines, or participants who are unwilling to modify their benzodiazepine use will.
* Pregnant or breastfeeding women will be excluded, as well as women of childbearing potential who will not use a medically acceptable method of contraception (i.e. IUD, oral contraceptives).
* Participants who are deaf, blind, or experience any other significant sensory impairment that would preclude them from completing study procedures will also be excluded, as well as participants who are unable to understand study procedures or provide informed consent.
* Participants receiving isoniazid or ethionamide, or who have a known sensitivity to D-cycloserine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A. Eden Evins, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital - Center For Addiction Medicine, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One hundred fifty participants were enrolled (signed consent), but only 98 were found eligible and started study procedures. Eighty one participants started smoking cessation CBT, and 62 finished and were randomized to receive either D-cycloserine or identical placebo added to exposure treatment to prevent relapse to smoking.
Pre-assignment Details: Participants received their choice of nicotine patch or varenicline (0.5 mg per day for 3 days, 0.5 mg bid for 4 days, 1 mg bid for 4 wks) and weekly cognitive behavioral therapy for smoking cessation.
Groups:
- Placebo: 50 mg capsule,single dose, twice, one week apart, by mouth
  Placebo
Period: Overall Study
Arm/Group | Placebo | D-cycloserine
Started | 32 | 30
Completed | 28 | 28
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Population: After 4 wks of smoking cessation treatment and CBT, participants who had 18 hrs of abstinence, smoking no cigarettes for at least 18 hrs and CO<10ppm were randomized
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | D-cycloserine | Total
Number analyzed (Participants) | 32 | 30 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (11.4) | 48.4 (12.4) | 47.7 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 22 | 41
  Male | 13 | 8 | 21

OUTCOME MEASURES:

1. Primary Outcome: Effect of D-cycloserine + Cue-exposure Treatment on Continuous Abstinence From Tobacco Smoking.
Description: Participants assigned to receive D-cycloserine + CET will achieve better maintenance of tobacco abstinence, as assessed with self-report and saliva cotinine measurements, than those who receive placebo + CET at week 6 follow up visits
Time Frame: Up to 6 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | D-cycloserine
Number analyzed (Participants) | 32 | 30
percentage of participants | 9 | 30

2. Secondary Outcome: Effect of D-cycloserine + Cue-exposure Treatment on Skin Conductance
Description: Recently abstinent smokers assigned to receive D-cycloserine + CET will have less physiologic (skin conductance) reactivity to smoking cues at the Post-Extinction Assessment than those who receive placebo + CET.
  Subjects were presented with 2 blocks of audio recordings, one smoking-related script and one neutral script unrelated to smoking. Assessment of skin conductance was made after each audio recording was presented. The skin conductance mean was obtained for each script (smoking vs neutral). Differences in responsivity (skin conductance) to smoking cues (smoking script) was compared between subjects who received D-cycloserine + CET and subjects who received placebo + CET.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: change in microSiemens
Arm/Group | Placebo | D-cycloserine
Number analyzed (Participants) | 32 | 30
change in microSiemens | 0.14 (0.46) | 0.18 (0.31)
Statistical Analysis 1: Comparison: Placebo vs D-cycloserine; Test type: Superiority; p = 0.574, ANOVA
Statistical Analysis 2: Comparison: Placebo vs D-cycloserine; Test type: Superiority; p = 0.747, ANOVA

3. Secondary Outcome: Effect of D-cycloserine + Cue-exposure Treatment on Heart Rate
Description: Recently abstinent smokers assigned to receive D-cycloserine + CET will have less physiologic (heart rate) reactivity to smoking cues at the Post-Extinction Assessment than those who receive placebo + CET.
  Subjects were presented with 2 blocks of audio recordings, one smoking-related script and one neutral script unrelated to smoking. Heart rate measurement was obtained after each audio recording was presented. The heart rate mean was obtained for each script (smoking vs neutral). Differences in responsivity (heart rate) to smoking cues (smoking script) was compared between subjects who received D-cycloserine + CET and subjects who received placebo + CET.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: change in beats per minute
Arm/Group | Placebo | D-cycloserine
Number analyzed (Participants) | 32 | 30
change in beats per minute | -0.13 (2.64) | 0.98 (2.34)
Statistical Analysis 1: Comparison: Placebo vs D-cycloserine; Test type: Superiority; p = 0.94, ANOVA

4. Secondary Outcome: Effect of D-cycloserine + Cue-exposure Treatment on Electromyogram
Description: Recently abstinent smokers assigned to receive D-cycloserine + CET will have less physiologic (electromyogram) reactivity to smoking cues at the Post-Extinction Assessment than those who receive placebo + CET.
  Subjects were presented with 2 blocks of audio recordings, one smoking-related script and one neutral script unrelated to smoking. Electromyogram of the corrugator (EMGc)measurement was obtained after each audio recording was presented. The EMGc mean was obtained for each script (smoking vs neutral). Differences in responsivity (EMGc) to smoking cues (smoking script) was compared between subjects who received D-cycloserine + CET and subjects who received placebo + CET.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: change in micro volts
Arm/Group | Placebo | D-cycloserine
Number analyzed (Participants) | 32 | 30
change in micro volts | 0.25 (1.02) | 0.46 (1.52)
Statistical Analysis 1: Comparison: Placebo vs D-cycloserine; Test type: Superiority; p = 0.818, ANOVA

5. Secondary Outcome: Effect of D-cycloserine + Cue-exposure Treatment on Craving
Description: Recently abstinent smokers assigned to receive D-cycloserine + CET will have less craving at the Post-Extinction Assessment than those who receive placebo + CET The scale used to measure craving was a Visual Analogue Scale 0 (no desire at all) - 7 (unable to resist) Subjects were presented with 2 blocks of audio recordings, one smoking-related script and one neutral script unrelated to smoking. Craving level was obtained after each audio recording was presented. The craving mean was obtained for each script (smoking vs neutral). Differences in craving level response to smoking cues (smoking script) was compared between subjects who received D-cycloserine + CET and subjects who received placebo + CET.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: change in units on a scale
Arm/Group | Placebo | D-cycloserine
Number analyzed (Participants) | 32 | 30
change in units on a scale | 2.28 (2.30) | 1.44 (1.87)
Statistical Analysis 1: Comparison: Placebo vs D-cycloserine; Test type: Superiority; p = 0.123, ANOVA

6. Secondary Outcome: Effect of D-cycloserine + Cue-exposure Treatment on Attentional Bias Toward Smoking Cuesmeasured With the Emotional Stroop Task
Description: Recently abstinent smokers assigned to receive D-cycloserine + CET will have less attentional bias (Smoking Stroop task) toward smoking cues at the Post-Extinction Assessment than those who receive placebo + CET The Emotional Stroop uses smoking-related words and neutral words to measure attentional bias toward smoking related cues. Attentional bias is a central feature of many cognitive theories of addiction and can be measured with an emotional analog of the Stroop task. In this task, participants name the colors in which words are printed, and the words vary in their relevance to smoking. Extensive research has shown that patients are often slower to name the color of a word associated with concerns relevant to their clinical condition due to distraction by the meaning of the word(Williams, Mathews et al. 1996). The Stroop interference Score is obtained by subtracting Reaction Time (RT) to smoking minus the Reaction Time to neutral
Time Frame: Baseline and week 6
Measure: Mean (Standard Deviation); unit: Stroop interference Score
Arm/Group | Placebo | D-cycloserine
Number analyzed (Participants) | 32 | 30
Stroop interference Score | 35.27 (74.93) | 50.30 (74.85)
Statistical Analysis 1: Comparison: Placebo vs D-cycloserine; Test type: Superiority; p = 0.473, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Placebo | D-cycloserine
Serious Adverse Events (participants affected / at risk) | 1/32 | 0/30
Other Adverse Events (participants affected / at risk) | 24/32 | 24/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=32) | D-cycloserine (N=30)
compression fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=32) | D-cycloserine (N=30)
Anorexia (General disorders) | 2 | 4
Blurred vision (General disorders) | 3 | 3
Constipation (Gastrointestinal disorders) | 6 | 6
Depressen mood (Psychiatric disorders) | 9 | 9
Diarrhea (Gastrointestinal disorders) | 9 | 2
Dizziness (General disorders) | 3 | 4
Dry mouth (General disorders) | 9 | 7
Enuresis (General disorders) | 3 | 2
Fever (General disorders) | 2 | 1
Headache (General disorders) | 4 | 3
Hypersalivation (General disorders) | 2 | 2
Insomnia (General disorders) | 8 | 7
Irritability (Psychiatric disorders) | 11 | 9
Malaise (General disorders) | 7 | 4
Nausea (Gastrointestinal disorders) | 5 | 2
Skin rash (Skin and subcutaneous tissue disorders) | 5 | 4
Restlessness (Psychiatric disorders) | 2 | 7
Drowsiness (General disorders) | 6 | 5
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Stiffness (General disorders) | 3 | 4
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 5
Vomiting (Gastrointestinal disorders) | 2 | 2
Other (General disorders) | 14 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No